CLINICAL TRIAL: NCT03643848
Title: Sleep-dependent Negative Overgeneralization in Peri-pubertal Anxiety
Brief Title: Sleep and Emotional Memory in Peripubertal Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R01MH116005-01 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-08-23 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: Per NIMH policy at the time of funding, the current trial is considered a clinical trial due to prospective, randomized assignment to an "intervention" to observe effects on behavioral or health related outcomes. The "intervention" for Aim 3 (n=60) includes randomized assignment to sham sounds (sounds unrelated to the memory task) or target sounds (sounds that were played during the time of the memory task) that are played during sleep to cue memory processing.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind (participant, outcome assessor) for Aim 3 (sham versus target sounds)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep with Sound Cues (Experimental): Sounds played at time of memory encoding will be replayed during sleep to cue memory processing.
  Interventions: Behavioral: Sleep with Sound Cues
- Sleep with Sham Cues (Sham Comparator): Sounds that were not played at time of memory encoding will be played during sleep as a sham comparison
  Interventions: Behavioral: Sleep with Sham Cues

INTERVENTIONS:
Behavioral: Sleep with Sound Cues — Experimental manipulation to observe effects on memory for learned material.
  Arms: Sleep with Sound Cues
Behavioral: Sleep with Sham Cues — Sham manipulation
  Arms: Sleep with Sham Cues

SUMMARY:
The current study aims to deepen understanding of the symptom dimension of negative overgeneralization in anxiety. Specifically, the study examines the malleability of memory processes that are known to occur during sleep that may underlie negative overgeneralization.

DETAILED DESCRIPTION:
Up to 50% of peripubertal youth with anxiety have unmet clinical needs, leaving these youth at high risk for suicide, depression and substance abuse across adolescence. In accord with the NIMH strategic plan, the proposal aims to deepen mechanistic understanding of anxiety during the sensitive period of peripuberty to inform novel treatments and reduce health risks. The focus is on negative overgeneralization, which is a core dimension of anxiety that is poorly understood, and refers to the tendency to generalize aversive responses from one context (house fire) to other contexts (camp-fire) that share features. Amygdala activity, induced by heightened emotional arousal, enhances plasticity in associative learning mechanisms, facilitating the binding of contextual features in memory that are only loosely related. The proposal posits that sleep plays a critical role in negative overgeneralization. Specifically, the proposal draws from basic neuroscience to posit a model by which heightened amygdala reactivity during wakefulness, induced by increased emotional arousal, facilitates replay of negative memories during sleep. This facilitated replay leads to the stabilization and integration (consolidation) of negative memories into long-term memory networks via slow wave oscillatory events during NREM sleep. The proposal further posits that facilitated replay of negative memories during sleep promotes generalization by influencing underlying neurocomputational mechanisms (i.e., pattern completion - a computational process that makes neural representations similar). Finally, the proposal posits that sleep-dependent consolidation is malleable, such that Targeted Memory Reactivation (TMR) of positive memories during sleep can competitively displace consolidation of negative memories. This model is tested using a novel multi-method approach combining neuroimaging, polysomnography, and a memory task that captures behavioral generalization and its underlying neural mechanisms (i.e. pattern completion).

Aims 1 and 2 do not involve a clinical trial. Aim 1 examines 200 peripubertal youth (ages 10-13 years) across a full continuum of anxious symptoms in a randomized sleep (n=140) versus wake (n=60) design to demonstrate sleep-dependent effects on behavioral and neural mechanisms of negative overgeneralization. Aim 2 focuses on the 140 youth in the sleep condition to evaluate amygdala reactivity at encoding and sleep neurophysiology during post-encoding sleep as mediators between anxiety and negative overgeneralization.

Aim 3 is the clinical trial to which this registration refers. In Aim 3, the same design as the sleep condition (above) is used, but a new sample of youth with elevated anxiety (n=60) is recruited to enroll in a randomized trial in which neutral memories are cued during sleep (TMR, n=30), or sham cues are presented during sleep (n=30), to examine malleability of sleep-dependent mechanisms of negative overgeneralization. This project will set the stage for the long-term goal of developing novel interventions that manipulate sleep (e.g. via TMR) not only to improve existing symptoms, but also to positively shape neurodevelopment and reduce risk in the sensitive period of peripuberty.

ELIGIBILITY:
Inclusion Criteria:

* 10-13 years old
* Able to understand and communicate in English and have a parent who is able to understand and communicate in English or Spanish
* included across any range of symptoms of anxiety, and may meet full diagnostic criteria for Social Phobia, Generalized Anxiety and Separation Anxiety.
* be right-handed.

Exclusion Criteria:

* For youth to be excluded from participation, they must:

(A) meet diagnostic criteria for Organic Mental Disorders, Psychotic Disorders, Pervasive Developmental Disorders (including autism spectrum disorders), Obsessive Compulsive Disorder, Attention-Deficit Hyperactivity Disorder, Conduct Disorder, Oppositional Defiant Disorder, Posttraumatic Stress Disorder, Bipolar Disorder, Tic disorder, Impulse Control Disorder, or Intellectual Disability. However, to improve generalizability, if Attention-Deficit Hyperactivity Disorder, Oppositional Defiant Disorder, Obsessive Compulsive Disorder, Mood Disorders (including past or present episodes of Major Depressive Disorder and/or dysthymia) or Posttraumatic stress Disorder co-occurs with an anxiety disorder (see Inclusion Criteria above) participants may be included.

(B) Children complete the Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-II). Scores below 80 (i.e., two standard deviations below normed mean) are considered exclusionary for this study.

(C) show high likelihood and/or serious intent of hurting themselves or others.

(D) have not been living with a primary caregiver for at least 6 months who is legally able to give consent for the child's participation.

(E) be a victim of previously undisclosed abuse requiring investigation or ongoing supervision by the Department of Children and Families;

(F) have a serious vision problem that is not corrected with prescription lenses, or have prescription glasses outside of the range of -5.00 to +3.00 (contact lenses are ok).

(G) have a physical disability that interferes with their ability to lie in scanner and/or click a mouse button rapidly;

(H) have a serious hearing problem;

(I) have a history of neurological or other major medical conditions affecting brain function.

(J) current or past history of sleep disorder, as assessed during the screening; exclusionary sleep disorders will include sleep apnea, and circadian rhythm disturbances (i.e., advanced or delayed sleep-phase)

(K) self-reported average sleep duration < 6 hours or > 11 hours across weekday and weekend nights, or normal bedtime later than 1:00 am; .

(L) Are not suitable to undergo MRI scanning due to claustrophobia, certain implanted devices/metal (e.g., cardiac pacemaker, neurostimulator, some artificial joints, metal pins, surgical/aneurysm clips, heart valves, cochlear implants, retinal implants, shrapnel in eye, non-removable body piercing or other non-MRI compatible metal/device.

(M) Are pregnant.

(N) Some Color Tattoos.

(O) Color Contacts.

(P) Currently sick or recovering from illness.

(Q) Currently taking non-stimulant psychotropic medications. However, participants who have been off non- stimulant medication for at least 2 weeks (the typical washout period) may be included. Participants currently taking stimulant medications may be included, as long as medication was not taken within 24 hours of scans (at the discretion of the parent/legal guardian and prescribing physician).

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana McMakin, PhD, Principal Investigator — Florida International University and Nicklaus Children's Hospital; Aaron Mattfeld, PhD, Principal Investigator — Florida International University
Locations (2):
- United States (2):
  - Center for Children and Families, Florida International University, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
yes, data are shared via NIH NDA and include behavioral, imaging, polysomnography and clinical data.
Supporting Information: Study Protocol, SAP
Time Frame: supporting docs available as part of original NIH grant. We will share individual data via NIH NDA per NIH policy timelines and guidance.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment from community and outpatient mental health clinics for children
Period: Overall Study
Arm/Group | Sleep With Sound Cues | Sleep With Sham Cues
Started | 29 | 29
Completed | 28 | 28
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep With Sound Cues | Sleep With Sham Cues | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants] — Range= 10.0-13.11 years
  Participants
    <=18 years | 29 | 29 | 58
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Range=10.0-13.11 years
  years | 11.4 (1.1) | 11.4 (1.1) | 11.4 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 22 | 43
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 21 | 22 | 43
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 1 | 1
Anxiety Severity Composite [Mean (Standard Deviation); unit: units on a scale (standardized factor)] — The Composite Anxiety Score is a continuous score derived from a principal components analysis (PCA) across multiple anxiety-report items from youth (Scared scale), caregiver (Scared scale), and clinician (PARS-6; ADIS diagnosis) informants. It is designed to capture a latent trait anxiety factor that integrates information across measures. Values range from-0.45 (lowest anxiety) to +3.9 (highest anxiety).
  Higher scores = greater anxiety severity/worse outcome; Lower scores = lower anxiety severity/better outcome.
  units on a scale (standardized factor) | 1.4 (1.0) | 1.3 (1.2) | 1.4 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Scores on the Lure Generalization Index (a Behavioral Measure of Generalization)
Description: Emotional Mnemonic Similarity Task. Participants view pictures depicting negative or neutral objects/scenes. After a delay period (1 week) they are presented with a second set of pictures that are the same (targets), slightly different (lures), or completely different (foils) from the first series of pictures. They are told to indicate by button press if images they are currently viewing are "old" or "new". Responding to the lures as old ("false alarms") provides a signature of generalization for each participant. To correct for response biases (i.e., a tendency to label items as "old") a Lure Generalization Index (LGI) is calculated which reflects corrected memory generalization by subtracting false alarm rates to foils from false alarm rates to lures. Larger LGI values indicate greater generalization (i.e., greater tendency to misidentify similar items as previously seen, accounting for overall biases to identify any items as previously seen). Minimum value -1 and maximum value =1
Time Frame: Delayed recall, 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sleep With Sound Cues (Targeted Memory Reactivation [TMR]): Sounds played at time of memory encoding for neutral stimuli will be replayed during sleep to cue neutral memory processing (and displace negative memory processing).
  Sleep with Sound Cues: Experimental manipulation to observe effects on memory for learned material.
- Sleep With Sham Cues (Sham): Sounds that were not played at time of memory encoding will be played during sleep as a sham comparison
  Sleep with Sham Cues: Sham manipulation
Arm/Group | Sleep With Sound Cues (Targeted Memory Reactivation [TMR]) | Sleep With Sham Cues (Sham)
Number analyzed (Participants) | 28 | 28
units on a scale
  Lure Generalization Index for Negatively Valenced Stimuli | .24 (.16) | .26 (.12)
  Lure Generalization Index for Neutral Stimuli | .14 (.15) | .10 (.11)
Statistical Analysis 1: Comparison: Sleep With Sound Cues (Targeted Memory Reactivation [TMR]) vs Sleep With Sham Cues (Sham); Condition (TMR, Sham) x Valence (Negative, Neutral) predicting Lure Generalization Index at 1 week. We hypothesized a significant interaction, with a reduction in negative generalization and an increase in neutral generalization in the TMR condition; Test type: Superiority; p < .046, Mixed Models Analysis — a priori threshold p<.05; REML; Satterwaite method for t-tests.Participant is random effect. Addtnl fixed effects: Valence, Condition, Anxiety Severity, Gender, Age (months); variance components; inferring mean diff = 0.068, Standard Deviation .033

2. Secondary Outcome: Scores on the Lure Generalization Index (a Behavioral Measure of Generalization)
Description: Emotional Mnemonic Similarity Task. Participants view pictures depicting negative or neutral objects/scenes. After a delay period (12 hours) they are presented with a second set of pictures that are the same (targets), slightly different (lures), or completely different (foils) from the first series of pictures. They are told to indicate by button press if images they are currently viewing are "old" or "new". Responding to the lures as old ("false alarms") provides a signature of generalization for each participant. To correct for response biases (i.e., a tendency to label items as "old") a Lure Generalization Index (LGI) is calculated which reflects corrected memory generalization by subtracting false alarm rates to foils from false alarm rates to lures. Larger LGI values indicate greater generalization (i.e., greater tendency to misidentify similar items as previously seen, accounting for overall biases to identify any items as previously seen). Minimum value -1 and maximum value =1
Time Frame: Recall, 12 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sleep With Sound Cues (Targeted Memory Reactivation [TMR]): Sounds played at time of memory encoding of neutral stimuli will be replayed during sleep to cue memory processing of neutral stimuli (and displace processing of negative stimuli).
  Sleep with Sound Cues: Experimental manipulation to observe effects on memory for learned material.
Arm/Group | Sleep With Sound Cues (Targeted Memory Reactivation [TMR]) | Sleep With Sham Cues (Sham)
Number analyzed (Participants) | 29 | 29
units on a scale
  Lure Generalization Index for Negatively Valenced Stimuli | .40 (.19) | .40 (.21)
  Lure Generalization Index for Neutral Stimuli | .26 (.19) | .30 (.16)
Statistical Analysis 1: Comparison: Sleep With Sound Cues (Targeted Memory Reactivation [TMR]) vs Sleep With Sham Cues (Sham); Condition (TMR, Sham) x Valence (Negative, Neutral) predicting Lure Generalization Index at 12 hour test. We hypothesized a significant interaction, with a reduction in negative generalization and an increase in neutral generalization in the TMR condition; Test type: Superiority; p = .61, Mixed Models Analysis — a priori p<.05; included additional fixed effects: Anxiety severity, gender, age (months); variance components; inferring mean diff = -.033, Standard Error of Mean .064

ADVERSE EVENTS:
Time Frame: From consent through study completion, which was approximately 2 weeks after the experimental manipulation (or "intervention"). For the two participants who did not complete the study, they were monitored until their withdrawal.
Description: Participants at risk for Serious Adverse Events, All-Cause Mortality and Other Adverse Events is N=58
Arm/Group | Sleep With Sound Cues | Sleep With Sham Cues
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
Pilot study--small sample size, should be interpreted with caution until replication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03643848/Prot_SAP_000.pdf